CLINICAL TRIAL: NCT05969704
Title: Magnetic Resonance Imaging Targeted (fusion) Versus Cognitive Prostatic Biopsy in Biopsy-naïve Suspected Cancer Prostate Patient a Comparison Study
Brief Title: Fusion Versus Cognitive MRI Targeted Prostatic Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Shebl Mehanna, Doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TRUS prostatic biopsy
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Cancer
Keywords: fusion biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fusion biopsy (Active Comparator): This biopsy procedure that combines the pictures from an MRI and an ultrasound to create a detailed 3-D image of the prostate. This procedure makes it easier to see an abnormal area of prostate in order to guide the biopsy needle into the abnormal area. A sample of tissue can then be taken and checked under a microscope for cancer. A fusion biopsy may help find prostate cancer cells that may be missed with other types of biopsies. It may help find cancer at an early stage and plan cancer treatment.
  Interventions: Procedure: MRI fusion targeted prostatic biopsy
- cognitive biopsy (Active Comparator): the biopsy operator reviews the MR images and creates a mental three-dimensional representation of the prostate and of the lesion within it to take a biopsy from it
  Interventions: Procedure: MRI cognitive targeted prostatic biopsy

INTERVENTIONS:
Procedure: MRI fusion targeted prostatic biopsy — combines the pictures from an MRI and an ultrasound to create a detailed 3-D image of the prostate. This procedure makes it easier to see an abnormal lesion of prostate in order to guide the biopsy needle into the abnormal lesion
  Other Names: fusion biopsy
  Arms: fusion biopsy
Procedure: MRI cognitive targeted prostatic biopsy — the biopsy operator reviews the MR images and creates a mental three-dimensional representation of the prostate and of the lesion within it to take a biopsy from the lesion
  Other Names: cognitive biposy
  Arms: cognitive biopsy

SUMMARY:
The aim of the present study is to compare the accuracy of Magnetic resonance imaging targeted (fusion) versus cognitive prostatic biopsy in biopsy-naïve suspected cancer prostate patient

DETAILED DESCRIPTION:
Prostate cancer is the second most frequent malignancy (after lung cancer) in men worldwide, counting 1,276,106 new cases and causing 358,989 deaths (3.8% of all deaths caused by cancer in men.

The clinical prostate cancer detection rate of TRUS-guided needle biopsies is only 25-30%. while more than 50% of cancers that require definitive treatment remain undetected during initial biopsies .

Clinical studies have shown that 75-80% of non-palpable carcinomas remain undetected during initial prostate biopsies.

Multi-parametric prostate MRI has a high sensitivity for the detection of prostate adenocarcinoma and has shown promise for targeted biopsy of lesions that may be missed on routine systematic trans -rectal ultrasound (TRUS) biopsy .

The most recent European Association of Urology guidelines recommend MRI before prostate biopsy for biopsy-naïve men with elevated PSA, the strength rating of the recommendation is weak.

A systematic 12-core trans-rectal ultrasound-guided systematic biopsy (TRUS-SB) is still carried out for biopsy-naïve men at present. However, the TRUS-SB technique has several limitations, including over-diagnosis of clinically insignificant prostate cancer (CISCa), under-diagnosis of clinically significant prostate cancer (CSCa), false negative biopsy results and biopsy-related complications, such as bleeding and infections .

Targeted prostate biopsies from MRI-suspicious lesions have been shown to improve the cancer detection rate (CDR) of CSCa compared with systematic TRUS-guided biopsies .

Currently, three biopsy techniques are used for TB from MRI-suspicious lesions: in-bore MRI biopsies, cognitive magnetic resonance imaging trans-rectal ultrasound fusion targeted biopsy (COG-TB) and software guided magnetic resonance imaging-ultrasound fusion targeted biopsies (MRUS-TB). Inbore MRI biopsies that are carried out with an MRI-compatible guidance device can target suspicious lesions accurately; however, such biopsies are time-consuming and expensive .

In the COG-TB technique, a physician samples a location that has been visually estimated using ultrasound and is considered to correspond to the location of a suspicious lesion that was detected on MRI. However, when the suspicious lesion is completely invisible (isoechoic or too small) on TRUS, the accuracy of such biopsies is likely reduced .

The accuracy of COG-TB might be influenced by multiple factors, including the alignment of prostate landmarks, the physician's experience and so on. for these reasons, MRUS-TB where software fuses the MRI images with real-time TRUS images to guide the operator to biopsy the suspicious lesions is more commonly carried out; however, the optimal TB method remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* prostate biopsy-naïve men
* PSA levels of up to 20 ng/mL
* Multi-parametric prostate MRI revealed a PIRAD 4 or PIRAD 5.

Exclusion Criteria:

* PSA level greater than 20 ng/mL
* patient with history of TRUS biopsy
* patient diagnosed as cancer prostate or with distant metastasis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
detection of clinically significant prostate cancer | two weeks
  accuracy of MRI targeted fusion versus cognitive prostatic biopsy in biopsy-naïve suspected cancer prostate patient to detect clinically significant prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University Hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided